CLINICAL TRIAL: NCT00102193
Title: A Randomized, Prospective, Double-Blinded, Placebo-Controlled (Sham-Controlled) Study to Evaluate the Safety and Effectiveness of the Adacolumn Apheresis System for the Treatment of Moderate to Severe Ulcerative Colitis
Brief Title: Study for the Treatment of Ulcerative Colitis With Adacolumn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 512-04-205
Record Dates: First submitted 2005-01-24; First posted 2005-01-25 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis, Apheresis
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Device: Adacolumn Apheresis System

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the Adacolumn Apheresis System to treat the signs and symptoms of ulcerative colitis.

DETAILED DESCRIPTION:
Trial Features:

* Non-drug therapy
* Most patients can remain on current treatment regimen, including prednisone, budesonide and medications such as Asacol (mesalamine), Pentasa (mesalamine), Colazal (balsalazide disodium) and Dipentum (olsalazine sodium) throughout the study

Components of the Study:

* Study length is 24 weeks, which includes a screening visit, ten treatment visits over nine weeks and 4 follow-up appointments
* Physical exams, laboratory tests and disease assessments conducted at no charge to the patient
* 2:1 Randomization (treatment:sham)

ELIGIBILITY:
Key Inclusion Criteria:

* Moderate to severe active ulcerative colitis with colonic involvement with ulcerative colitis beyond 15 cm of the anal verge
* Adequate peripheral venous access to allow for completion of the apheresis treatments
* Receiving one or more of the following medical therapies:

  *sulfasalazine, *mesalamine and other 5-ASA agents, *prednisone or 6-mercaptopurine or azathioprine OR Have not received the above medical therapies due to intolerance or demonstrated non-response
* Agree to participate in the required follow-up visits
* Able to complete a diary
* Signed written informed consent document and authorization for use of protected health information

Key Exclusion Criteria:

* Evidence of toxic megacolon
* Major surgery within the past 6 weeks or anticipated need for surgery within 12 weeks
* Proctocolectomy, total colectomy, ileostomy, stoma or ileal pouch-anal anastomosis
* Requiring in-patient hospitalization
* A history of allergic reaction to heparin or heparin-induced thrombocytopenia
* A history of hypersensitivity reaction associated with an apheresis procedure or intolerance of apheresis procedures
* A history of severe cardiovascular or peripheral arterial diseases
* A history of cerebral vascular diseases
* Liver diseases
* Renal insufficiency
* Insulin-dependent Type I or Type II diabetes
* Known bleeding disorder or use of concomitant anticoagulant therapy for purposes other than apheresis treatment
* Any hypercoagulable disorder
* Known infection with Hepatitis B or C, or HIV
* Severe anemia
* Leukopenia or granulocytopenia
* Evidence of current systemic infection
* Malignancy
* Pregnant, lactating or planning to become pregnant during the course of the investigational study
* Used within the last 30 days, an investigational drug, biologic or device or 5 half-lives, if known, for any investigational drug or biologic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168
Dates: Start 2004-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness will be primarily evaluated at Week 12 by disease activity index (DAI) score
Safety will be evaluated by determining the frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yosuke Komatsu, MD, PhD, Study Director — Otsuka America Pharmaceutical
Locations (37):
- United States (26):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - Providence Clinical Research, Burbank, California
  - University of California, San Francisco, San Francisco, California
  - Rocky Mountain Gastroenterology Associates, PC, Wheat Ridge, Colorado
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago, Department of Medicine, Section of Gastroenterology, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Massachusetts General Hospital, GI Unit, Boston, Massachusetts
  - Tufts University School of Medicine, Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Clinton Township, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Long Island Clinical Research Associates, Great Neck, New York
  - University of North Carolina, Division of Digestive Disease & Nutrition, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Digestive Disease Specialists Inc., Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
- Canada (11):
  - Walter Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Gastroenterology and Hepatology Clinic, Abbotsford, British Columbia
  - St Paul's Hospital, University of British Columbia, Vancouver, British Columbia
  - Hotel-Dieu Hospital, Kingston, Ontario
  - London Health Sciences Centre, South Street Campus, London, Ontario
  - London Health Sciences Centre, University Campus, London, Ontario
  - The Ottawa Hospital-Civic Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec